CLINICAL TRIAL: NCT04206202
Title: Application of 3D Printing Patient-specific Instrumentation in Total Knee Arthroplasty
Brief Title: 3D Printing Guides in Total Knee Arthroplasty
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Southwest Hospital, China (Other)
Responsible Party: Principal Investigator, Xiaojun Duan, Deputy Director of the Center for Joint Surgery, Southwest Hospital, China
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 3DKneeGuide
Record Dates: First submitted 2019-12-15; First posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Osteoarthritis of the Knee
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PSI group (Experimental): 3D-printed patient-specific instrumentation (PSI) will be used in the total knee arthroplasty (TKA) of this group.
  Interventions: Device: 3D-Printed Patient-Specific Intramedullary Guide

INTERVENTIONS:
Device: 3D-Printed Patient-Specific Intramedullary Guide — The 3D-printed patient-specific intramedullary guide is used in TKA to control femoral component rotation.

SUMMARY:
This study aims to design a patient-specific instrumentation to be used in total knee arthroplasty and evaluate its accuracy of femoral component rotation and intramedullary guide so as to explore its clinical effects.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is the most universal and effective means for treating terminal stage osteoarthritis (OA) of knee. With the development of three-dimensional printing (3DP) technology in the medical domain, the application of patient-specific instrumentation (PSI) in arthroplasty has become more common. The aim of this study was to design a PSI to achieve appropriate femoral resection and accurate component rotation for a successful TKA, and to explore its clinical effects.

ELIGIBILITY:
Inclusion Criteria:

* Patients with advanced OA of the knee, varus deformity of no more than 15 degrees, flexion-contracture deformity of no more than 10 degrees, without extra-articular deformity of the knee;
* Weight-bearing radiograph of the X-ray image showed the OA Kellgren-Lawrence classification grade Ⅳ;
* The treatment for the patient was TKA, whether or not to use PSI depends on the actual grouping.

Exclusion Criteria:

* Patients with varus deformity of more than 15 degrees, flexion-contracture deformity of more than 10 degrees of the knee;
* Patients with traumatic arthritis and inflammatory arthritis;
* Patients with huge bone defects around the knee
* Patients who had active infection around the knee;
* Patients with knee valgus deformity;
* Patients with severe extra-articular deformity;
* Patients who had previous knee surgery;
* Patients who had periarticular soft tissue dysfunction and neuropathy;
* Patients who had poor physical condition and could not withstand the operation;
* Patients who refused to be followed.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-05-01 (Actual); Primary Completion 2020-03-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of the radiological outcomes | Postoperative 12 months
  The radiological outcomes include the hip-knee-ankle angle (HKA), posterior condylar angle (PCA), patella transverse axis-femoral transepicondylar axis angle (PFA) of the patients. The data were collected to evaluate the accuracy of the 3DP-designed PSI.

SECONDARY OUTCOMES:
Hospital for Special Surgery knee score (HSS) | Postoperative 1,6,12 months
  Hospital for Special Surgery knee score (HSS) was used to evaluate postoperative recovery of knee function in an adult population. The HSS score system mainly includes 6 aspects as pain, function, muscle force, deformity, stability, and the range of motion. The score standard had a maximum of 100 points (best possible outcome). A total score <60 is considered a poor score, 60-69 fair,70-85 is good and 86-100 excellent.
American Knee Society knee score (AKS) | Postoperative 1,6,12 months
  The AKS was used to evaluate postoperative recovery of knee function in an adult population. The HSS score system mainly includes 4 aspects as pain, stability, range of motion and the function. The score standard had a maximum of 100 points (best possible outcome). A total score <60 is considered a poor score, 60-69 fair,70-85 is good and 86-100 excellent.

CONTACTS AND LOCATIONS:
Overall Officials: Rui He, M.D., Principal Investigator — Southwest Hospital, China
Locations (1):
- Southwest Hospital, Chongqing, China